CLINICAL TRIAL: NCT06967766
Title: A Complex Intervention to Promote Appropriate Antibiotic Use Among Rural Residents Based on the Metaphor-Embedded Integrated Behavioral Model
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bo Yan (Other)
Responsible Party: Sponsor-Investigator, Bo Yan, Doctor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ZGL202504-10
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Antimicrobial Drug Resistance
Keywords: health education; Metaphor
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metaphor-based health education (Experimental): In each intervention scenario, health education information is set to target key behaviors in the scenario. In the main scenarios for obtaining antibiotics, such as township health centers, village clinics, and community pharmacies, scenario-driven interventions are carried out for two key behaviors: patients actively asking for antibiotics (led by doctors in township health centers) and customers buying antibiotics without prescriptions (led by community pharmacy staff).
  Interventions: Behavioral: health education based on the Metaphor-Embedded Integrated Behavioral Model
- Regular education (No Intervention)

INTERVENTIONS:
Behavioral: health education based on the Metaphor-Embedded Integrated Behavioral Model — In each intervention scenario, health education information is set to target key behaviors in the scenario. In the main scenarios for obtaining antibiotics, such as township health centers, village clinics, and community pharmacies, scenario-driven interventions are carried out for two key behaviors: patients actively asking for antibiotics (led by doctors in township health centers) and customers buying antibiotics without prescriptions (led by community pharmacy staff).
  Arms: Metaphor-based health education

SUMMARY:
The study aims to address the question of how to provide effective health education on health topics with high medical specialisation (e.g. bacterial drug resistance in this study), especially for rural or low-educated populations. In response to the high degree of correlation between irrational antimicrobial drug use behaviours, how to achieve the effectiveness of interventions on the complex health topic of rational use of antimicrobial drugs through synergistic interventions with multiple scenarios?

In this study, the investigators used an experimental-like research design to conduct a full-scenario intervention involving antimicrobial drug acquisition, use, and disposal in a township-based approach, so as to reduce the prevalence of irrational antimicrobial drug use behaviours among rural residents, and to significantly improve the governance of antimicrobial drug use in rural areas. After six months of intervention, the following specific objectives were achieved:

1. The incidence of self-treatment and use of antimicrobial drugs in the intervention group decreased by 30% compared with the control group;
2. Rational use of antimicrobial drugs and awareness of bacterial drug resistance among rural residents in the intervention group increased by 50% compared with the control group;
3. In the intervention group, the incidence of rural residents actively asking for antimicrobial drugs when seeking medical treatment, actively purchasing antimicrobial drugs without prescription at community pharmacies, stocking up on antimicrobial drugs at home, and improperly disposing of antimicrobial drugs decreased by 40%, 30%, 30%, and 50%, respectively, compared with that of the control group.

The study included the development and testing of metaphorical health materials and a multi-contextual metaphorical health education intervention. The implementation of the intervention included training in metaphorical health education and doctor-patient communication, a multi-situational intervention based on the theory of metaphorically embedded integrative behaviours, and the design of incentives for standardised antimicrobial drug discarding.

ELIGIBILITY:
Inclusion Criteria:

* Residents aged 18 years and over who have lived in the survey township for more than 6 months

Exclusion Criteria:

* Residents with mental illness, severe mental health problems, and those unable to complete the questionnaire

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
antibiotic use | six months
  Changes in antibiotic use rates among sick rural residents in the past month(self-treatment with antibiotics and antibiotics prescribed by doctors when seeking medical treatment)

SECONDARY OUTCOMES:
knowledge | six months
  Rational use of antibiotics and awareness of bacterial resistance among rural residents
Prevalence of unsolicited requests for antimicrobial drugs at medical appointments | six months
  Question：Did you voluntarily ask your doctor for antibiotics during your visit? The options contain yes and no.
Prevalence of unsolicited purchase of antimicrobials without a prescription at a pharmacy | six months
  Question：In the past month, have you gone to the pharmacy and voluntarily purchased antibiotics without a doctor's prescription? Options include yes and no.
Proportion of residents stocking antimicrobial drugs at home | six months
  Do you currently keep antibiotics in your home? (Do not include antibiotics that have been prescribed for you or a family member by your doctor and that you are currently taking) The options include yes, no and unknown.
Incidence of unregulated disposal of antimicrobial drugs | six months
  Questions：
  1. Have you disposed of antibiotics that you no longer use in your home?
  2. If yes, how did you handle it the last 1 time? The options include ①Throw it into the rubbish bin ②Pour it into a flush toilet or sink and flush it away ③Give it to someone else ④Send it to a pharmacy/medical institution, etc. for recycling ⑤Recycle it through electronic platforms such as Alipay ⑥ Give it to a professional for disposal ⑦ Other (please specify)